CLINICAL TRIAL: NCT00834990
Title: A Relative Bioavailability Study of 500 mg Divalproex Sodium Delayed-Release Tablets Under Non-Fasting Conditions
Brief Title: Divalproex Sodium Delayed-Release Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R03-593
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: divalproex sodium
- 2 (Active Comparator)
  Interventions: Drug: Depakote®

INTERVENTIONS:
Drug: divalproex sodium — delayed-release 500 mg tablet
  Arms: 1
Drug: Depakote® — delayed-release 500 mg tablet
  Arms: 2

SUMMARY:
This study will compare the relative bioavailability of 500 mg Divalproex Sodium Delayed-Release Tablets with that of 500 mg Depakote® Tablets following a single oral dose (1 x 500 mg tablets) in healthy subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Screening Demographics: All subjects selected for this study will be healthy men or women 18-65 years of age, inclusive, at the time of dosing. The subject's body mass index (BMI) should be less than or equal to 30.
* Screening Procedures: Each subject will complete the screening process within 28 days prior to period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed and signed by each potential participant before full implementation of screening procedures.

Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.

The screening clinical laboratory procedures will include:

* HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count
* CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase
* HIV antibody, hepatitis B surface antigen, hepatitis C antibody screens
* URINALYSIS: by dipstick; full microscopic examination if dipstick positive
* URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine
* SERUM PREGNANCY SCREEN (female subjects only)
* FOLLICLE STIMULATING HORMONE (FSH; female subjects only): verify postmenopausal status

If female and:

* Is postmenopausal for at least 1 year with postmenopausal status defined as: > 60 years of age and amenorrheic for at least one year; if 60 years of age or younger, must also have a serum FSH level > 30 IU/L; or
* Is surgically sterile for at least 6 months (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria

* Subjects with a recent history of drug or alcohol addiction or abuse.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a positive hepatitis B surface antigen screen, a positive hepatitis C antibody screen, or a reactive HIV antibody screen.
* Subjects demonstrating a positive drug abuse screen when screened for this study.
* Female subjects demonstrating a positive pregnancy screen.
* Female subjects who are currently breastfeeding.
* Subjects with a history of allergic response(s) to divalproex sodium or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Subjects who currently or report using tobacco products within 90 days of Period I dose administration.
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Subjects who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Subjects who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 28 days prior to Period I dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to Period I dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute
Locations (1):
- PRACS Institute Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Divalproex Sodium First: 500 mg Divalproex Sodium Delayed Release Tablets test product dosed in first period followed by 500 mg Depakote® Delayed Release Tablets reference product dosed in the second period.
- Depakote® First: 500 mg Depakote® Delayed Release Tablets reference product dosed in first period followed by 500 mg Divalproex Sodium Delayed Release Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Divalproex Sodium First | Depakote® First
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Divalproex Sodium First | Depakote® First
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Divalproex Sodium First | Depakote® First
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Divalproex Sodium First | Depakote® First | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1 | 0 | 1
  White | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Divalproex Sodium: 500 mg Divalproex Sodium Delayed Release Tablets test product dosed in either period.
- Depakote®: 500 mg Depakote® Delayed Release Tablets reference product dosed in either period.
Arm/Group | Divalproex Sodium | Depakote®
Number analyzed (Participants) | 23 | 23
µg/mL | 49.02 (7.61) | 47.83 (9.57)
Statistical Analysis 1: Comparison: Divalproex Sodium vs Depakote®; Test type: Non-Inferiority or Equivalence — The pharmacokinetic parameters were evaluated statistically by an analysis of variance (ANOVA) appropriate for the experimental design of this study; Ratio of the T/R geometric mean x 100 = 103.41, 90% CI [97.13 to 110.08] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Divalproex Sodium | Depakote®
Number analyzed (Participants) | 23 | 23
µg*h/mL | 934.87 (193.26) | 917.11 (192.97)
Statistical Analysis 1: Comparison: Divalproex Sodium vs Depakote®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101.68, 90% CI [96.79 to 106.83] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Divalproex Sodium | Depakote®
Number analyzed (Participants) | 23 | 23
µg*h/mL | 1024.72 (223.2) | 991.74 (224)
Statistical Analysis 1: Comparison: Divalproex Sodium vs Depakote®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 103.17, 90% CI [98.5 to 108.05] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.